CLINICAL TRIAL: NCT06860243
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of MK-5684 in Male Participants With Moderate Hepatic Impairment
Brief Title: A Study to Evaluate Opevesostat (MK-5684) in Male Participants With Moderate Hepatic Impairment (MK-5684-009)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 5684-009; MK-5684-009 (Other: MSD)
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hepatic Impairment; Healthy Participants
MeSH Terms: interventions — Prednisone; fludrocortisone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moderate Hepatic Impairment (Experimental): On Day 1, participants with moderate hepatic impairment will receive a single oral dose of opevesostat under fasting conditions and a single dose of hormone replacement therapy (HRT) (prednisone and fludrocortisone acetate) under fed conditions approximately 4.5 hours after opevesostat dosing. Participants with moderate hepatic impairment will receive another dose of HRT on Day 2.
  Interventions: Drug: Opevesostat; Drug: Prednisone; Drug: Fludrocortisone acetate
- Healthy (Experimental): On Day 1, healthy participants will receive a single oral dose of opevesostat under fasting conditions and a single dose of HRT (prednisone and fludrocortisone acetate) under fed conditions approximately 4.5 hours after opevesostat dosing.
  Interventions: Drug: Opevesostat; Drug: Prednisone; Drug: Fludrocortisone acetate

INTERVENTIONS:
Drug: Opevesostat — Oral film-coated tablet
  Other Names: MK-5684
Drug: Prednisone — Oral tablet
Drug: Fludrocortisone acetate — Oral tablet

SUMMARY:
Researchers have designed a study medicine called opevesostat as a new way to treat prostate cancer.

The purpose of this study is to learn what happens to opevesostat in a person's body over time (a pharmacokinetic [PK] study). Researchers will compare what happens to opevesostat in the body when it is given to healthy participants and participants with moderate hepatic (liver) impairment.

ELIGIBILITY:
The main inclusion criteria include but are not limited to the following:

* All participants:
* Is a continuous non-smoker or moderate smoker (≤ 10 cigarettes per day or equivalent) for at least 3 months prior to dosing
* Has body mass index (BMI) ≥ 18.0 and ≤ 42.0 kg/m2
* Participants with moderate hepatic impairment:
* Has a diagnosis of chronic, stable, hepatic insufficiency with features of cirrhosis due to any etiology

The main exclusion criteria include but are not limited to the following:

* All participants:
* Has a first-degree relative with multiple unexplained syncopal events, unexplained cardiac arrest, or sudden cardiac death, or has a known family history of an inherited arrhythmia syndrome (including Brugada syndrome)
* Has a history of cancer (malignancy)
* Has positive results for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Participants with moderate hepatic impairment
* Has unstable electrolyte abnormalities or electrolyte abnormalities that are considered difficult to manage for participants with hepatic impairment
* Has a history of liver or other solid organ transplantation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-02-09 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration Versus Time Curve from 0 to Infinity (AUC0-inf) of Opevesestat | At designated timepoints (up to approximately 96 hours post-dose)
  Plasma samples will be collected to determine the AUC0-inf of opevesostat.
Area Under the Concentration Versus Time Curve from 0 to the Last Quantifiable Sample (AUC0-last) of Opevesestat | At designated timepoints (up to approximately 96 hours post-dose)
  Plasma samples will be collected to determine the AUC0-last of opevesostat.
Area Under the Concentration Versus Time Curve from 0 to 24 hours (AUC0-24) of Opevesestat | At designated timepoints (up to approximately 24 hours post-dose)
  Plasma samples will be collected to determine the AUC0-24 of opevesostat.
Maximum Observed Concentration (Cmax) of Opevesestat | At designated timepoints (up to approximately 96 hours post-dose)
  Plasma samples will be collected to determine the Cmax of opevesostat.
Time to Maximum Concentration (Tmax) of Opevesestat | At designated timepoints (up to approximately 96 hours post-dose)
  Plasma samples will be collected to determine the Tmax of opevesostat.
Apparent Terminal Half-life (t1/2) of Opevesestat | At designated timepoints (up to approximately 96 hours post-dose)
  Plasma samples will be collected to determine the t1/2 of opevesostat.
Apparent Clearance (CL/F) of Opevesestat | At designated timepoints (up to approximately 96 hours post-dose)
  Plasma samples will be collected to determine the CL/F of opevesostat.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of Opevesestat | At designated timepoints (up to approximately 96 hours post-dose)
  Plasma samples will be collected to determine the Vz/F of opevesostat.

SECONDARY OUTCOMES:
Number of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 2 weeks
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 2 weeks
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami ( Site 0002), Miami, Florida
  - Texas Liver Institute ( Site 0001), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/